CLINICAL TRIAL: NCT03247153
Title: Influence of Corticosteroid Therapy on Heart Function
Brief Title: Influence of Corticosteroids on Heart Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HYMC-52-17
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Heart; Complications
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corticosteroid Therapy Patients (Experimental): Corticosteroid therapy patients will be examined by echocardiography before, during and after receiving treatment
  Interventions: Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Echocardiography — Imaging of the heart using ultrasound

SUMMARY:
This study will examine the effect of corticosteroid treatment on heart function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with good echogenic body structure
* Patients with sinus rhythm with no conduction disorder

Exclusion Criteria:

* Patients with major medical condition
* Patients who are not hemodynamical stable
* Patients receiving long-term corticosteroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Changes in heart function | One month after completion of treatment
  Comparison of echocardiography performed before, during, and after corticosteroid administration will display changes in heart function

CONTACTS AND LOCATIONS:
Overall Officials: Nina Avshovitch, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No